CLINICAL TRIAL: NCT05861947
Title: A Phase I, Open Label, Dose-Escalation, First in Human (FIH) Study Evaluating the Safety, Pharmacokinetics, Pharmacodynamics and Efficacy of AUR106 in Patients With Select Relapsed Advanced Malignancies (JIVAN)
Brief Title: A Phase 1 Clinical Trial of AUR106 in Patients With Relapsed Advanced Malignancies
Acronym: JIVAN
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aurigene Discovery Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AUR106-101
Record Dates: First submitted 2023-04-25; First posted 2023-05-17 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-04

CONDITIONS: Relapse; Advanced Malignant Neoplasm; Non Small Cell Lung Cancer; Gastric Cancer; Urothelial Carcinoma; Kidney Cancer; Colon Cancer; Esophagus Cancer
MeSH Terms: conditions — Recurrence; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Carcinoma, Transitional Cell; Kidney Neoplasms; Colonic Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose Escalation "3+3" Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AUR106 (Experimental): 25mg to 100 mg, Currently planned dose levels are 25 mg QD, 50 mg QD, 25 mg BID, 50 mg BID, 100 mg BID
  Interventions: Drug: AUR106

INTERVENTIONS:
Drug: AUR106 — Once or twice daily

SUMMARY:
A Phase I, Open Label, Dose-Escalation, First in Human (FIH) Study Evaluating the Safety, Pharmacokinetics, Pharmacodynamics and Efficacy of AUR106 in Patients with Select Relapsed Advanced Malignancies (JIVAN).

DETAILED DESCRIPTION:
This is a Phase I, Open Label, Dose-Escalation, First in Human (FIH) study in adult patients with select relapsed advanced malignancies. The safety and tolerability of oral AUR106 will be evaluated in patients with selected advanced solid tumors (Non-small cell lung cancer, Gastric cancer, Urothelial cancer, Kidney cancer, Colon cancer and Esophageal cancer), who do not have any available curative or life prolonging treatment options and have exhausted all effective locally available therapies. The traditional 3+3 design for dose escalation will be used to evaluate safety, PK/PD and determine the Optimal Biological Dose (OBD) of AUR106, as a single agent. The Optimal Biological Dose will be selected using a totality of safety, PK and PD data.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated informed consent and agree to comply with all study related activities.
2. Male or female patients aged ≥ 18 years.
3. Patients have to meet the following criteria:

   * Pathological diagnosis of the following solid tumors: Non-small cell lung cancer, Gastric cancer, Urothelial cancer (includes bladder cancer and cancers of ureter / renal pelvis), Kidney cancer, Colon cancer, Esophageal cancer).
   * Standard curative or life prolonging measures do not exist, and patient must have exhausted all effective therapies, available locally. At a minimum, patients should have received at least 2 lines of therapy in the metastatic setting.
   * Standard treatment options provided to the patients are exhausted.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Patients with disease related ECOG 2 are allowed, in addition to ECOG 0 and 1).
5. Acceptable bone marrow as described below:

   * ANC ≥ 1500/μL (without WBC growth factor support).
   * Platelet count ≥ 100,000/μL without transfusion support.
   * Hemoglobin ≥ 9 g/dL (Transfusion is allowed to achieve this Hb).
6. Acceptable organ function as described below:

   * Total Bilirubin ≤ 1.5 x ULN (Patients with known Gilbert's syndrome are allowed with a Total Bilirubin ≤ 2.5 x ULN).
   * AST (SGOT) ≤ 3 x ULN (≤ 5 × ULN if known liver metastases).
   * ALT (SGPT) ≤ 3 x ULN (≤ 5 × ULN if known liver metastases).
   * Creatinine clearance (CrCl) ≥ 60 mL/min (either measured or estimated by the Cockcroft-Gault formula). (Cockcroft-Gault formula for estimated creatinine clearance [eCrCl]: eCrCl = [140 - Age] × Weight [kg] × [0.85 if Female] / [72 × serum creatinine (mg/dL)]).
   * Albumin ≥ 3.0 g/dL.
7. Ability to swallow and retain oral medications.
8. Negative serum pregnancy test in women of childbearing potential (WOCBP).
9. Women of childbearing potential and men who partner with such a woman of childbearing potential must agree to use one or more of highly effective method(s) of contraception for the duration of the study, i.e., through 28-day follow up visit, after discontinuation of study drug(s).
10. Evidence of measurable disease per RECIST, v1.1 for solid tumors (Eisenhauer et al. 2009). Measurable disease for solid tumors is defined as at least one lesion that can be accurately measured in at least 1 dimension with a minimum size of 10 mm for non-nodal lesions or 15 mm in short axis for nodal lesions.

Exclusion Criteria:

1. Systemic anti-cancer therapy, such as chemotherapy, biological therapy, or immunomodulatory drug therapy, received within the past 28 days or 5 half-lives, whichever is longer, from the Cycle 1 Day 1 of the study.
2. Presence of an acute or chronic toxicity resulting from prior anti-cancer treatment, with the exception of alopecia or nail changes, that has not resolved to Grade ≤ 1, as determined by NCI CTCAE v 5.0.
3. Definitive Radiotherapy within the last 21 days of Cycle 1 Day 1 (limited field palliative radiation is allowed and no restrictions during the screening period or during the trial).
4. Use of any investigational agent within 28 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
5. Known symptomatic or untreated or recently treated (≤ 6 months of screening) central nervous system (CNS) metastases. Patients with previously treated (> 6 months of screening) and are now stable and asymptomatic, from CNS perspective, are allowed.
6. Major surgery ≤ 28 days from Cycle 1 Day 1 (major surgery is defined as a procedure requiring general anesthesia).
7. Known to be human immunodeficiency virus (HIV) positive or have an acquired immunodeficiency syndrome-related illness.
8. Known active or chronic hepatitis B or hepatitis C infection.
9. Uncontrolled congestive heart failure (New York Heart Association [NYHA] Class 2-4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to Cycle 1 Day 1.
10. Ongoing cardiac dysrhythmias requiring treatment of any grade or treatment of cardiac dysrhythmias in past 3 months, before Cycle 1 Day 1.
11. The QTcF (corrected QT interval Fridericia method) value in the screening ECG > 460 ms in both males and females.
12. Previous or concomitant additional malignancy, except for basal-cell or squamous cell carcinoma of the skin or carcinoma-in-situ of the uterine cervix; patients with other malignancies are eligible if they have remained disease free for at least 2 years prior to trial entry and in the opinion of the investigator deemed to have a low likelihood of recurrence.
13. Pregnant or lactating women.
14. Any clinically significant medical, psychiatric or social condition; or laboratory abnormality that may increase the risk of trial participation or may interfere with the informed consent process and/or with compliance with the requirements of the trial or may interfere with the interpretation of the trial results and, in the Investigator's opinion, would make the patient inappropriate for entry into this trial.
15. Patients who require concomitant administration of drugs which have a high risk of prolonging QT interval.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-26 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Optimal Biological Dose (OBD) | First 28 Days (Cycle 1)
  To determine the Optimal Biological Dose (OBD) based on safety, pharmacokinetic, and pharmacodynamic data
Dose Limiting Toxicity (DLT) | First 28 Days (Cycle 1)
  To determine the DLT of AUR106
Pharmacokinetics: Area under the curve (AUC) | Day 1 and Day 15
  Area under the curve of AUR106
Pharmacokinetics: Maximum concentration Pharmacokinetics: Maximum concentration | Day 1 and Day 15
  Maximum concentration of AUR106
Pharmacokinetics: Time to Maximum concentration | Day 1 and Day 15
  Time to Maximum concentration of AUR106
Pharmacokinetics: Terminal elimination half life | Day 1 and Day 15
  Terminal elimination half life of AUR106

SECONDARY OUTCOMES:
Adverse Events | Through study completion, an average of 1 year
  Adverse Events as characterized by type, frequency, severity (as per CTCAE Version 5.0), timing, seriousness, and relationship to study therapy.
Laboratory abnormalities | Through study completion, an average of 1 year
  Number of participants with abnormal laboratory tests results

OTHER OUTCOMES:
Exploratory endpoint (PD biomarker): CD3 level | Day 1, Day 8 and Day 15
  Change in CD3 level
Exploratory endpoint (PD biomarker): CD4 level | Day 1, Day 8 and Day 15
  Change in CD4 level
Exploratory endpoint (PD biomarker): CD8 level | Day 1, Day 8 and Day 15
  Change in CD8 level
Exploratory endpoint (PD biomarker): CD56 level | Day 1, Day 8 and Day 15
  Change in CD56 level
Exploratory endpoint (PD biomarker): IL-2 level | Day 1, Day 8 and Day 15
  Change in IL-2 level
Exploratory endpoint (PD biomarker): IL-6 level | Day 1, Day 8 and Day 15
  Change in IL-6 level
Exploratory endpoint (PD biomarker): IFN-γ level | Day 1, Day 8 and Day 15
  Change in IFN-γ level

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Kumar, MD, Study Director — Head Clinical Development
Locations (6):
- India (6):
  - Omega Hospital, Visakhapatnam, Andhra Pradesh
  - Unique Hospital Multispeciality and Research Institute, Surat, Gujarat
  - Kiran Multi Super Specialty Hospital, Surat, Gujarat
  - Sankalp Speciality Hospital, Nashik, Maharashtra
  - Moraya Multispeciality Hospital (Ashwin Medical Foundations), Pune, Maharasthra
  - All India Institute of Medical Sciences, Bhubaneswar, Odisha

IPD SHARING:
Plan to Share IPD: No